CLINICAL TRIAL: NCT01059136
Title: Aldosterone Lethal Effects Blocked in AMI Treated With or Without Reperfusion to Improve Outcome and Survival at Six Months Follow-up: THE ALBATROSS TRIAL
Brief Title: Aldosterone Blockade Early After Acute Myocardial Infarction
Acronym: ALBATROSS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P071216
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Outcome; Aldosterone; Spironolactone
MeSH Terms: conditions — Myocardial Infarction | interventions — Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1:Spironolactone (Experimental): Aldosterone blockade on top of standard therapy
  Interventions: Drug: Spironolactone
- 2:Standard therapy (No Intervention): Standard therapy

INTERVENTIONS:
Drug: Spironolactone — Unique 200mg IV dose of Potassium Canrenoate followed by 25 mg daily oral dose of Spironolactone for 6 months
  Arms: 1:Spironolactone

SUMMARY:
Study hypothesis : An early blockade of aldosterone receptors initiated at the first medical contact after acute myocardial infarction may reduce major cardiovascular events within 6 months after the occurrence of the myocardial infarction.

Primary efficacy criterion : The 6 month rate of the composite of death, resuscitated cardiac arrest, potentially lethal ventricular arrhythmia, indication for implantation of an implantable cardioversion device, occurrence or aggravation of heart failure.

Primary objective: To demonstrate the superiority of aldosterone blockade initiated as soon as possible within 72 hours after the onset of acute myocardial infarction on top of standard therapy, compared to standard therapy alone, with or without reperfusion therapy.

Study design : Prospective, multi-centre randomised, open labeled with 2 parallel study arms.

DETAILED DESCRIPTION:
Rational :The blockade of the renin-angiotensin-aldosterone (RAA) pathway by angiotensin conversion enzyme inhibitors (ACEI) is one corner stone in the management of heart failure as well as the management of ischemic heart disease, especially after acute myocardial infarctionHigh plasma aldosterone levels have been associated with both direct and indirect toxic effects on myocardium. ACEIs are associated with partial and temporary reduction of plasma aldosterone levels.The RALES randomized controlled trial has shown a reduction of mortality associated with the use of the selective aldosterone receptor blocker spironolactone, on top of standard therapy including ACEIs in the setting of NYHA 3-4 chronic heart failure. The EPHESUS randomized controlled trial has shown a reduction of mortality associated with the use of another selective aldosterone receptor blocker Eplerenone, initiated 3 to 14 days after acute myocardial infarction complicated by clinical heart failure and left ventricular ejection fraction < 40%.Both previous studies have also reported a rapid reduction of global and arrhythmia-related mortality, within 30 days after the initiation of the medication.Such benefit has been reported after delayed initiation of aldosterone blocked, while aldosterone is at its highest level at presentation after acute myocardial infarction, with a rapid decrease within days after admission. Furthermore high aldosterone levels on admission are associated with adverse outcome independent of heart failure.

The ALBATROSS trial :Hypothesis: An early blockade of aldosterone receptors initiated at the first medical contact after acute myocardial infarction may reduce major cardiovascular events within 6 months after the occurrence of the myocardial infarction.

Primary objective: To demonstrate the superiority of aldosterone blockade initiated as soon as possible within 72 hours after the onset of acute myocardial infarction on top of standard therapy, compared to standard therapy alone, with or without reperfusion therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 ans
2. Ischemic symptom of ≥ 20 minutes
3. Randomization within 72 hours after symptom onset
4. Electrocardiogram or biological evidence of myocardial infarction:

   * ST segment elevation ≥ 2 mm in ≥ 2 adjacent precordial derivations
   * ST segment elevation ≥ 1 mm in ≥ 2 adjacent peripheral derivations
   * New left bundle branch block
   * New significant Q wave in ≥ 2 adjacent peripheral derivations
   * Troponin levels ≥3 times upper local limit of normal values and Thrombolysis In Myocardial Infarction (TIMI) non-ST elevation myocardial infarction risk score ≥ 3.
5. Patients with health insurance
6. Written informed consent obtained from:

   1. - the patient
   2. -A member of the family or the person of confidence if the patient is unable to provide informed consent

Exclusion Criteria:

1. Contraindication or known intolerance to study drugs
2. Patients already treated by aldosterone blockers for diseases other than systemic hypertension (e.g. primary hyperaldosteronism)
3. Hyperkaliemia >5.5 mmol/l at the time of randomization
4. Renal function impairment :Plasma creatinin level > 220 µmol/l and/or Creatinin clearance 30 ml/min
5. Severe liver deficiency (Child-Pugh Class 3)
6. Pregnant or breast feeding women, or women desiring pregnancy within 6 months after randomization
7. Patients already included in another biomedical intervention trial
8. Life expectancy < 1 year
9. Cardiac arrest lasting (ECM) >10 minutes prior to randomization
10. Patient unable or unwilling to comply with the treatment or the follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1603 (Actual)
Dates: Start 2010-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The 6 month rate of the composite of death, resuscitated cardiac arrest, potentially lethal ventricular arrhythmia, indication for implantable cardioversion device, occurrence or aggravation of heart failure. | 6 months

SECONDARY OUTCOMES:
Any of the criteria of the primary endpoint | 6 months
primary endpoint+ myocardial infarction+stroke cardiovascular death | 6 months
death + resuscitated cardiac arrest | 6 months
Death+resuscitated cardiac arrest+ventricular arrhythmia+indication for implantable defibrillator device | 6 months
death+heart failure | 6 months
Acute renal failure | 6 months
primary endpoint | hospital discharge and 30 days
rate of hyperkaliemia (> 5.5 mmol.l-1) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Farzin BEYGUI, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital PITIE-SALPETRIERE - Institut de Cardiologie, Paris, France

REFERENCES:
- [Derived] Hashimoto H, Yamada H, Murata M, Watanabe N. Diuretics for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2025 Jan 29;1(1):CD014937. doi: 10.1002/14651858.CD014937.pub2. PMID 39878152
- [Derived] Beygui F, Cayla G, Roule V, Roubille F, Delarche N, Silvain J, Van Belle E, Belle L, Galinier M, Motreff P, Cornillet L, Collet JP, Furber A, Goldstein P, Ecollan P, Legallois D, Lebon A, Rousseau H, Machecourt J, Zannad F, Vicaut E, Montalescot G; ALBATROSS Investigators. Early Aldosterone Blockade in Acute Myocardial Infarction: The ALBATROSS Randomized Clinical Trial. J Am Coll Cardiol. 2016 Apr 26;67(16):1917-27. doi: 10.1016/j.jacc.2016.02.033. PMID 27102506
- [Derived] Beygui F, Vicaut E, Ecollan P, Machecourt J, Van Belle E, Zannad F, Montalescot G. Rationale for an early aldosterone blockade in acute myocardial infarction and design of the ALBATROSS trial. Am Heart J. 2010 Oct;160(4):642-8. doi: 10.1016/j.ahj.2010.06.049. PMID 20934557